CLINICAL TRIAL: NCT01555515
Title: Safety and Efficacy of Sustained Erythropoietin Therapy of Anemia in End Stage Renal Disease (ESRD) Dialysis Patients Using EPODURE Biopump
Brief Title: Epodure Therapy of Anemia in End Stage Renal Disease on Dialysis With Epodure Skin Implant
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: New protocol to start with improved product
Sponsor: Medgenics Medical Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG-001-03
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2015-10

CONDITIONS: Anemia; End Stage Renal Disease
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPODURE Low dose (Experimental): EPODURE pump secreting hEPO 18-25 IU/kg/day
  Interventions: Procedure: implantation of autologous skin graft after ex-vivo treatment; Biological: Subcutan implantation of autologus skin graft after ex-vivo treatment

INTERVENTIONS:
Procedure: implantation of autologous skin graft after ex-vivo treatment — Subcutan implantation of autologous skin graft after ex-vivo treatment
Biological: Subcutan implantation of autologus skin graft after ex-vivo treatment — Subcutan implantation of autologus skin graft after ex-vivo treatment

SUMMARY:
In this End Stage Renal Disease (ESRD) patients who need Erythropoietin (epo) hormone will get it by a small implant of skin using their own skin, the implant will be treated in the laboratory and programmed to secrete Epo. The implant secretes the patients own epo minimizing the need for injections for a period of up to 6 months.

DETAILED DESCRIPTION:
This will be a Phase I-II, open-label, single-center, uncontrolled, tailored dose study. The trial will be conducted in Israel at the Tel Aviv Sourasky Medical Center.

Subjects will undergo similar study procedures and evaluations; however each patient will receive his or her own individually targeted dose of EPO delivered via EPODURE Biopumps. The targeted dose may vary between 20IU/kg/d to 65IU/kg/d based on each patient's weight, the historical average EPO amount administered and historical Hb levels including at least the 3 months prior to inclusion in the study. The objective is maintaining Hb levels within the target range of 10-12 g/dl.

ELIGIBILITY:
Inclusion Criteria:1.

1. Adult male or female subjects between 18 to 75 years of age at the time of screening visit.
2. Subject diagnosed with Anemia due to Chronic Renal Failure CKD stage 5 on dialysis treatment for at least 3 months. Hb < 12g/dL on 2 consecutive measures
3. Kt/V >1
4. INR not higher than 1.2
5. Subjects who are clinically stable.
6. Serum albumin > 3.5
7. Subjects with adequate iron stores (transferrin saturation > 20.0% and/or ferritin > 100 ng/ml).
8. Signed written informed consent to participate in the study.

Exclusion Criteria:

1. Uncontrolled hypertension (defined as diastolic blood pressure > 110 mmHg or systolic blood pressure > 180 mmHg during screening).
2. Subjects who receive oral anti-coagulation treatment (warfarin)
3. Subjects who receive Acetyl Salicylic Acid [(ASA), aspirin] above 325 mg/day or patients who receive ASA treatment between 100mg/d and 325 mg/d who cannot discontinue it for 1 week prior to each EPODURE procedure
4. Patients currently receiving injections of long-acting ESA's (Aranesp, Mircera, etc.)
5. Congestive heart failure (New York Heart Association functional class III or IV).
6. Grand mal seizures within 2 years of the screening visit.
7. Clinical evidence of severe hyperparathyroidism as defined by PTH levels of > 10 times the upper normal limits.
8. Major surgery within 12 weeks of the screening visit.
9. Systemic hematologic diseases (e.g., sickle cell anemia, myelodysplastic syndromes, hematologic malignancy, myeloma, hemolytic anemia).
10. Current systemic infection, active inflammatory disease, or malignancy under treatment.
11. Subjects known to have tested positive at any time in the past for antibodies to erythropoietic proteins.
12. Subject has history of malignancy within the past 2 years prior to the screening visit, with the exception of basal cell carcinoma.
13. Subjects with other concurrent severe and/or uncontrolled medical condition which could compromise participation in the study (i.e. active infection, uncontrolled diabetes, uncontrolled hypertension, congestive cardiac failure, unstable angina, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, uncompensated cirrhosis, active upper GI tract ulceration).
14. Subject is currently enrolled in, or has not yet completed a period of at least 30 days since ending other investigational device or drug trial(s).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Hg maintenance with in the range of 10-12 gr/dl for the duration of 6 month | 6 months
  A Phase I-II, open-label. The trial will be conducted in Israel at the Tel Aviv Sourasky Medical Center.
  Subjects will undergo similar study procedures and evaluations; however each patient will receive his or her own individually targeted dose of EPO delivered via EPODURE Biopumps. The targeted dose may vary between 20IU/kg/d to 65IU/kg/d based on each patient's weight, the historical average EPO amount administered and historical Hb levels including at least the 3 months prior to inclusion in the study. The objective is maintaining Hb levels within the target range of 10-12 g/dl.

SECONDARY OUTCOMES:
REDUCING THE AMOUNT OF EXOGENOUS EPO ADMINISTRATION | During the first 6 months of evaluation
  The biopumps are expected to secret sufficient Epo to support the Hb lebel in the desired range of 10-12 gr/dl

CONTACTS AND LOCATIONS:
Overall Officials: Doron Schwartz, Professor, Principal Investigator — Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
Early phase study.